CLINICAL TRIAL: NCT02841228
Title: Intensity-modulated Radiotherapy (IMRT) With Simultaneous Integrated Boost (SIB) Dose Escalation to the Gross Tumor Volume (GTV) With Concurrent Chemotherapy for Stage II/III Non-small Cell Lung Cancer (NSCLC)
Brief Title: Intensity-modulated Radiotherapy (IMRT) With Simultaneous Integrated Boost (SIB) for Inoperable Non-small-cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Hui Wang, Chief of thoracic radiation oncology department, Hunan Province Tumor Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIB-IMRT
Record Dates: First submitted 2016-07-05; First posted 2016-07-22 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: SIB-IMRT; NSCLC; Radiochemothearpy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy, Intensity-Modulated; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IMRT + SIB + Chemotherapy (Experimental): For all patients, the dose to the PTV will be kept constant at 60 Gy in 30 fractions at 2.0 Gy per fraction, SIBV will be kept constant at 72 Gy in 30 fractions at 2.4 Gy per fraction. Fractions given once a day, 5 times a week for six weeks. All patients will receive standard concurrent chemotherapy.
  Interventions: Radiation: IMRT + SIB + Chemotherapy

INTERVENTIONS:
Radiation: IMRT + SIB + Chemotherapy — For all patients, the dose to the PTV will be kept constant at 60 Gy in 30 fractions at 2.0 Gy per fraction , SIBV will be kept constant at 72 Gy in 30 fractions at 2.4 Gy per fraction. Fractions given once a day, 5 times a week for six weeks. All patients will receive standard concurrent chemotherapy.

SUMMARY:
Lung cancer is one of the most common cancer and the leading causes of cancer death in worldwide. Approximately 80% of NSCLC were inoperable. The prognosis of patients with LA-NSCLC remains disappointing. Investigators hypothesized that use of simultaneous integrated boost intensity modulated radiotherapy (SIB-IMRT) technology can safety increasing the radiation dose and benefit for inoperable NSCLC patients.

DETAILED DESCRIPTION:
Lung cancer is one of the most common cancer and the leading causes of cancer death in patients worldwide. Approximately 80% of NSCLC were inoperable. Concurrent chemo-radiation therapy (CCRT) is a standard treatment for locally advanced NSCLC who are not candidates for surgery. Nevertheless, the prognosis of patients with locally advanced NSCLC (LA-NSCLC) is still poor. Local control (LC) after CCRT is one of the most important prognostic factors. Local failure is common after standard-dose chemoradiation for NSCLC. Studies of stereotactic body radiation therapy (SBRT) have shown a steep dose response in treating early-stage lung cancer. Improving the total dose and shortening the overall treatment time may be effective for improving the LC rates. However, problems remain due to the toxicity to adjacent critical structures (e.g,lung,heart, esophagus), the target volumes usually limits the doses escalated that cannot be safely delivered by conventional radiotherapy techniques. In order to avoid the acute and late radiation toxicity of normal tissues, different dose prescriptions can be delivered to different target volumes in the same fraction, which deliver a higher dose to the Gross Tumor Volume (GTV) and a relatively lower dose to the subclinical disease. The technique is called simultaneous integrated boost intensity modulated radiotherapy (SIB-IMRT).

Investigators hypothesized that use of SIB-IMRT technology can safety increasing the radiation dose and benefit for inoperable NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed NSCLC, inoperable stages IIA-IIIB, according to American Joint Committee on Cancer （AJCC）Cancer Stage 7th
2. Performance status 0 to 2, ≤5% weight loss within the past 6 months
3. A forced expiratory volume at 1 second of ≥ 1 L
4. Life expectancy > 3 months
5. No invasion of large vessels, heart, esophagus, spinal cord.
6. Based on conformal treatment planning, the volume of lung at or exceeding 20 Gy (V20) must have been≤30%, the mean esophagus dose≤34 Gy, and the volume of esophagus exceeding 55 Gy (V55)≤30%
7. Tolerable and agree for Intensity-Modulated Radiation Therapy（IMRT） and concurrent chemoradiotherapy
8. Without severe other diseases
9. Informed consent

Exclusion Criteria:

1. Had received prior thoracic radiotherapy
2. Supraclavicular lymph node metastasis, pleural or pericardial effusions, and superior vena cava syndrome
3. Pregnant and lactating women
4. Serious complications
5. Other primary malignancies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | up to 12 months
  Progression free survival is defined as the time (in months) from the date of admission to the date of progression or last follow-up

SECONDARY OUTCOMES:
Treatment-related toxicities | up to 6 months
  To assess the pulmonary, oesophageal and cardiac grade 3 or 4 toxicity occurring up to 3 and 6 months after radiotherapy, according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Overall Response Rate (ORR) | up to 3 months
  ORR is defined as the proportion of participants with an overall response of complete response (CR) of any duration, partial response (PR) of any duration for a minimum of 3 months from start of treatment. Per RECIST, CR: disappearance of all target lesions, all non-target lesions, and no new lesion; PR: a >=30% decrease in the sum of the longest dimensions of the target lesions (TLs) taking as a reference the baseline sum, no unequivocal progression of non-TLs, and no new lesions; progressive disease (PD), a >=20% increase in TLs, clearly worsening of non-TLs, or emergence of new lesions; stable disease (SD): no change or small changes that do not meet previously given criteria for CR, PR or PD.
Overall survival (OS) | up to 36 months
  Overall survival is defined as the time (in months) from the date of admission to the date of death from any cause or last follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan province tumor pospital, Changsha, Hunan, China

REFERENCES:
- [Derived] Yang W, Zeng B, Qiu Y, Tan J, Xu S, Cai Y, Zhou Y, Liu Z, Luo J, Wang H. A Dosimetric Comparison of Dose Escalation with Simultaneous Integrated Boost for Locally Advanced Non-Small-Cell Lung Cancer. Biomed Res Int. 2017;2017:9736362. doi: 10.1155/2017/9736362. Epub 2017 May 28. PMID 28630876